CLINICAL TRIAL: NCT00151671
Title: Prospective, Randomized, Double Blind, Placebo-Controlled Study Evaluating the Effect of Oral Immune-Enhancing Nutritional Supplement on Hepatic Function After Liver Resection for Primary or Secondary Cancer on Cirrhosis or Liver Fibrosis
Brief Title: Effect of a Perioperative Oral Nutritional Supplementation on Patients Undergoing Hepatic Surgery for Liver Cancer
Acronym: IMPACT
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: insufficient enrollment rate
Sponsor: Rennes University Hospital (Other)
Collaborators: Ministry of Health, France (Other Government); Novartis (Industry)
Responsible Party: Direction of Clinical Research and Strategy, Rennes University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AFSSAPS 21541; PHRC/02-10; CIC0203/012
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2012-02-27 (Estimated); Status verified 2008-09

CONDITIONS: Liver Cancer; Hepatocellular Carcinoma; Cirrhosis; Liver Fibrosis
Keywords: Surgery; Liver Cancer; Cirrhosis; Nutrition
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular; Fibrosis; Liver Cirrhosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Perioperative Oral Nutritional Supplementation
  Interventions: Drug: Oral Impact®
- 2 (Placebo Comparator): Placebo of Perioperative Oral Nutritional Supplementation
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oral Impact® — Oral nutritional supplement containing L-arginin, ω3 polyunsaturated fatty acids, and nucleotides. Given three times a day for the 7 last preoperative and the first 3 postoperative days.
  Arms: 1
Drug: Placebo — Oral solution of placebo. Given three times a day for the 7 last preoperative and the first 3 postoperative days.
  Arms: 2

SUMMARY:
Cirrhotic patients undergoing hepatic resection have a mortality rate near 10%, and 30 to 70% of them develop severe complications. These failures are mainly due to hepatic insufficiency. Studies have already shown benefits of oral nutritional supplements in ORL, digestive, and cardiac surgery. We aimed to ascertain whether this nutritional, immune-enhancing supplementation, administered 7 days before and 3 days after surgery, could improve liver function and postoperative host defences in patients with liver cancer resection.

DETAILED DESCRIPTION:
In patients undergoing hepatic resection for liver cancer (with cirrhosis or fibrosis liver), mortality rate can reach 10% and morbidity (ascites, icteria, infections) 70%. These complications are mainly due to hepatic insufficiency: surgery leaves a reduced parenchyma, with oxidative stress lesions due to reperfusion injury. A good preoperative nutritional state has been shown to reduce complications and mortality. This can be amplified by preoperative nutrition with supplements containing L-arginin, ω3 polyunsaturated fatty acids, and nucleotides which boost immune responses, resistance to infections and liver function recovery. In this context, the study randomly assigns 50 patients who were scheduled to undergo hepatic resection, to receive either an oral immune-enhancing nutritional supplement or a placebo, for the 7 last preoperative and the first 3 postoperative days. The aim of the study is to evaluate the effects of this supplementation on liver function, immunity, and incidence of infections after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult over 18 years
* Hepatectomy of at least 2 segments
* For primary or secondary cancer
* With cirrhosis (Child Pugh <8) or liver fibrosis (fibrosis score of 3)
* Informed written consent

Exclusion Criteria:

* Pregnancy
* Recent weight loss of more than 10% of body weight
* Immunological deficiency
* Portal or hepatic arterial thrombosis
* Biliary duct dilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2003-04; Primary Completion 2008-04 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Factor V at day 3 after surgery | day 3

SECONDARY OUTCOMES:
Liver regeneration kinetics (bile production at days 1, 3, 5 and 7;factor V, γ-glutathione transferase, α-foetoprotein at days 1, 3, 5, 7, 10 and 30; liver volume at days 10 and 30 | days 1, 3, 5, 7, 10 and 30
Immunological biomarkers | Within 30 days
Infections | Within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Yannick Mallédant, MD, Study Director — Rennes University Hospital; Eric Bellissant, MD, PhD, Study Chair — Rennes University Hospital; Philippe Seguin, MD, Principal Investigator — Rennes University Hospital; Karim Boudjema, MD, PhD, Principal Investigator — Rennes University Hospital
Locations (1):
- Service de Réanimation Chirurgicale - Hôpital Pontchaillou, Rennes, France

REFERENCES:
- [Background] Tepaske R, Velthuis H, Oudemans-van Straaten HM, Heisterkamp SH, van Deventer SJ, Ince C, Eysman L, Kesecioglu J. Effect of preoperative oral immune-enhancing nutritional supplement on patients at high risk of infection after cardiac surgery: a randomised placebo-controlled trial. Lancet. 2001 Sep 1;358(9283):696-701. doi: 10.1016/s0140-6736(01)05836-6. PMID 11551575
- [Background] Senkal M, Zumtobel V, Bauer KH, Marpe B, Wolfram G, Frei A, Eickhoff U, Kemen M. Outcome and cost-effectiveness of perioperative enteral immunonutrition in patients undergoing elective upper gastrointestinal tract surgery: a prospective randomized study. Arch Surg. 1999 Dec;134(12):1309-16. doi: 10.1001/archsurg.134.12.1309. PMID 10593328
- [Background] Braga M, Gianotti L, Radaelli G, Vignali A, Mari G, Gentilini O, Di Carlo V. Perioperative immunonutrition in patients undergoing cancer surgery: results of a randomized double-blind phase 3 trial. Arch Surg. 1999 Apr;134(4):428-33. doi: 10.1001/archsurg.134.4.428. PMID 10199318